CLINICAL TRIAL: NCT06375408
Title: Clinical Study of Transcranial Alternating Current Stimulation in the Prevention of Delirium in Patients With Subarachnoid Hemorrhage
Brief Title: Transcranial Alternating Current Stimulation Prevents Delirium in Patients With Subarachnoid Hemorrhage
Acronym: TACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KS2022212
Record Dates: First submitted 2024-03-26; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-03

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid Hemorrhage; transcranial alternating current stimulation; delirium; Sleep quality
MeSH Terms: conditions — Subarachnoid Hemorrhage; Delirium; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The random number table method was used for randomization, and the envelope method was used for randomization. The random serial number was stored in an airtight envelope, an envelope was opened when a patient was admitted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group was treated with real transcranial alternating electrical stimulation.
  Interventions: Device: Real transcranial alternating electrical stimulation
- The control group (Sham Comparator): The control group was treated with sham transcranial alternating electrical stimulation.
  Interventions: Device: Sham transcranial alternating electrical stimulation

INTERVENTIONS:
Device: Real transcranial alternating electrical stimulation — The patients in the intervention group were treated with real tACS produced by Nexalin company. There were 3 treatment sites. According to the international 10-20 EEG system positioning method, one electrode was placed in the prefrontal lobe (Fp1, Fpz, Fp2 area, electrode size was 4.45cm×9.53cm), and the other two electrodes were placed in the left and right mastoid respectively (electrode size was 3.18cm×3.81cm). The treatment parameters were 40min twice daily with an interval of ≥4 hours for a total of 8 sessions over 4 days. tACS procedures were performed by trained and qualified full-time therapeutic nurses.
  Arms: The intervention group
Device: Sham transcranial alternating electrical stimulation — The patients in the control group were treated with sham tACS produced by Nexalin company. The fake tACS does not emit current, so it does not stimulate the cerebral cortex. The appearance, button, electrode, and quality of the fake tACS are exactly the same as those of the real tACS in patients' senses. There were 3 treatment sites. According to the international 10-20 EEG system positioning method, one electrode was placed in the prefrontal lobe (Fp1, Fpz, Fp2 area, electrode size was 4.45cm×9.53cm), and the other two electrodes were placed in the left and right mastoid respectively (electrode size was 3.18cm×3.81cm). The treatment parameters were 40min twice daily with an interval of ≥4 hours for a total of 8 sessions over 4 days. tACS procedures were performed by trained and qualified full-time therapeutic nurses.
  Arms: The control group

SUMMARY:
The goal of this clinical trial is to learn about using the latest transcranial alternating current stimulation (tACS) to reduce the incidence of delirium in patients with subarachnoid hemorrhage. The main question it aims to answer is:

• To evaluate the effect of tACS on reducing delirium in patients with subarachnoid hemorrhage.

Participants will treated with real tACS or sham tACS. Researchers will mainly compare the two groups to see if patients' delirium will reduce by using tACS.

DETAILED DESCRIPTION:
Research objectives: To reduce the incidence of delirium in patients with subarachnoid hemorrhage by using the latest transcranial alternating current stimulation.

Research contents:

1. To evaluate the effect of transcranial alternating current stimulation on improving sleep quality in patients with subarachnoid hemorrhage;
2. To evaluate the effect of transcranial alternating current stimulation on reducing delirium in patients with subarachnoid hemorrhage.

Research hypothesis: Transcranial alternating current stimulation can improve sleep quality and reduce the incidence of delirium in patients with subarachnoid hemorrhage.

Study design:

1. double-blind randomized clinical trial
2. Subjects：Patients with subarachnoid hemorrhage admitted to the neurosurgical intensive care unit during the study period.
3. Number of participating centers and names of centers: Single research center, Xuanwu Hospital, Beijing
4. Sample size: The total number of plans was 74, and the total number of study centers was 74.
5. Grouping of subjects：The random number table method was used for randomization, and the envelope method was used for randomization. The random serial number was stored in an airtight envelope, a patient was admitted, and an envelope was opened.
6. Intervention measures: ① The control group was treated with sham transcranial electrical stimulation; ② The experimental group was treated with real transcranial electrical stimulation.
7. Outcome measures: ① Efficacy indicators: the incidence and duration of delirium; The scores of Richard Campell sleep questionnaire, Hamilton Anxiety Scale, Mini-Mental State Examination, numerical rating scale for pain and muscle strength were recorded.② Safety indicators: the incidence of adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid hemorrhage was consistent with the Chinese Guidelines for the Diagnosis and Treatment of Subarachnoid Hemorrhage 2015;
* Patients after completion of surgical treatment;
* over 18 years of age;
* Hunt & Hess grade I-III;
* No major organ failure;
* The patient has no speech or hearing impairment;
* Informed consent of patients and their families, signed informed consent.

Exclusion Criteria:

* Those who have delirium at the time of enrollment;
* had substance abuse/dependence within 6 months before enrollment;
* had suffered from other mental illness within 6 months before enrollment;
* Suffering from serious or unstable organic diseases;
* Pregnant or lactating women and those planning to become pregnant in the near future;
* Damaged skin integrity at the electrode placement site, allergic to electrode gels or adhesives.
* with an implanted electronic stimulator;
* Patients who had received other noninvasive neuromodulation therapy within 1 month before enrollment;
* Participants in any other clinical trial within 1 month prior to baseline;
* There are circumstances in which the researcher considers it inappropriate to participate in this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium | up to 5days
  (occurrence of delirium was assessed 3 times a day from the start of the intervention to the day after the intervention ended ) Delirium incidence = Number of people who had experienced delirium within 5 days/total number of people in the intervention or control group.

SECONDARY OUTCOMES:
Sleep quality score | up to 5days
  The Richard Campell Sleep Questionnaire (RCSQ) consists of five sleep-related items: sleep depth, sleep fall, wake up during sleep, fall back to sleep, and overall sleep quality. A visual analog scale was used to score the patients, with each score ranging from 0 to 100. The average score of 5 sleep-related items was calculated, with 0 to 25 being low-quality sleep and 76 to 100 being high-quality sleep.
Anxiety score | up to 5days
  Hamilton Anxiety Scale (HAMA), which has 14 items, adopts a 5-level scoring method ranging from 0 to 4 points. The total score is the sum of the scores of 14 items, and the total score is >29 points, which may be severe anxiety. >21 points, there must be obvious anxiety; >14 points, there must be anxiety; More than 7 points, may have anxiety; If the score is less than 7, there is no anxiety symptom.
Duration of delirium | up to 5days
  The duration of patients' delirium from onset to end.
Cognitive function score | up to 5days
  mini-mental state examination (MMSE) : There are 30 items in the scale, each item is 1 point, one correct answer will get 1 point, the full score is 30 points, the higher the score, the better the cognitive function: MMSE≥27 is classified as normal, 21-26 as mild dementia, 10-20 as moderate dementia, and < 10 as severe dementia. MMSE is susceptible to the influence of education level, according to the level of education, its boundary standards are illiterate ≤17 points, primary school ≤20 points, secondary school or above education ≤24 points, indicating dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China